CLINICAL TRIAL: NCT01925469
Title: A Randomized Controlled Trial of Benzocaine Versus Placebo Spray for Pain Relief at Hysterosalpingogram
Brief Title: Benzocaine Versus Placebo Spray for Pain Relief at Hysterosalpingogram
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PFC-HSG-1
Record Dates: First submitted 2013-08-06; First posted 2013-08-19 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-03

CONDITIONS: Pain Relief; Analgesia
Keywords: Hysterosalpingogram; HSG; Pain relief; Analgesia; Benzocaine
MeSH Terms: conditions — Agnosia | interventions — Benzocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Benzocaine (Experimental): Benzocaine spray (14%), an FDA approved drug, will be used to assess whether this provides additional pain relief at time of hysterosalpingogram.
  Interventions: Drug: Benzocaine
- Saline spray (Placebo Comparator): A saline placebo spray will be used in the placebo group.
  Interventions: Drug: Saline spray

INTERVENTIONS:
Drug: Benzocaine
  Arms: Benzocaine
Drug: Saline spray — A saline spray will be used in the placebo group
  Arms: Saline spray

SUMMARY:
The objective of this study is to assess the utility of benzocaine spray versus a placebo spray in alleviating pain during and after hysterosalpingogram (HSG).

DETAILED DESCRIPTION:
Hysterosalpingography (HSG) is a radiographic evaluation during which a radio-opaque medium is inserted through the cervical canal in order to define the size and shape of the uterine cavity and patency of the fallopian tubes. The utility of HSG is an integral part of the evaluation of infertile women for intrauterine pathology. In some cases, HSG can be a painful procedure. Poor pain control can limit the quality of the study due to inability to complete the procedure in cases of extreme discomfort. There is little consensus regarding pain control during HSG, although a number of approaches have been studied. Patients undergoing HSG are typically advised to premedicate with ibuprofen, which is consistent with the current standard of care. This study will assess pain control using a benzocaine spray (in addition to ibuprofen) in patients undergoing routine HSG at the Hospital of the University of Pennsylvania. All patients who present to the Hospital of the University of Pennsylvania for HSG will be eligible for the study. Benzocaine spray versus a placebo spray will be applied to a tenaculum (a surgical hooklike instrument used to grasp and hold the cervix). The tenaculum will then be applied to the cervix prior to HSG and pain relief will be assessed at 3 time intervals: 0, 5, and 30 minutes. The primary outcome is the mean difference in patients pain score and will be measured using the Visual Analogue Scale (VAS) which has been shown to be a valid and reliable scale. The secondary outcome will assess patient satisfaction in each group using a validated patient satisfaction survey. The study design will be prospective, randomized, placebo controlled, and double blinded.

ELIGIBILITY:
Inclusion Criteria:

* All women who present to Penn Fertility Care over the age of 18 years old

Exclusion Criteria:

* Patients under the age of 18
* Pregnant patients
* Patients with a history of hypersensitivity to benzocaine
* Patients with a history of asthma or bronchitis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suleena K Kalra, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Bachman EA, Senapati S, Sammel MD, Kalra SK. Randomized controlled trial of benzocaine versus placebo spray for pain relief at hysterosalpingogram. Reprod Biomed Online. 2014 Jun;28(6):748-52. doi: 10.1016/j.rbmo.2014.02.012. Epub 2014 Mar 4. PMID 24745839

RESULTS

PARTICIPANT FLOW:
Groups:
- Benzocaine: Benzocaine spray (14%), an FDA approved drug, will be used to assess whether this provides additional pain relief at time of hysterosalpingogram.
  Benzocaine
Period: Overall Study
Arm/Group | Benzocaine | Saline Spray
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Benzocaine | Saline Spray | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (4.8) | 33.3 (6.5) | 33.9 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 8 | 6 | 14
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Nulliparous [Number; unit: participants] — A woman who has never had a child.
  participants | 12 | 12 | 24
Nulligravid [Number; unit: participants] — A woman who has never been pregnant
  participants | 7 | 10 | 17
History of dysmenorrhea [Number; unit: participants] | 7 | 6 | 13
History of chronic pelvic pain [Number; unit: participants] | 2 | 2 | 4
Pre-medication [Number; unit: participants] — "Pre-medication" includes ibuprofen or tylenol taken by patient prior to procedure.
  participants | 15 | 13 | 28
Bilateral obstruction [Number; unit: participants] | 2 | 1 | 3
Unilateral obstruction [Number; unit: participants] | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Score
Description: The primary outcome is the difference in pain score using a validated visual analog scale before the procedure, which is designated as the pre-procedure (or baseline) pain score to the maximum pain during procedure (designated as time 0) These two pain scores will be subtracted and the change in pain score will be reported. The validated visual analog scale allows patients to report pain on a scale of 0 to 100 mm long. At the beginning and at the end, there are two descriptors representing extremes of pain (i.e. no pain = 0 and extreme pain = 100). The patient rated her pain by making a vertical mark on the 100-mm line. The measurement in millimeters was converted to the same number of points ranging from 0 to 100 points. There are no subgroups.
Time Frame: Pre-procedure (Baseline) and procedure (Time 0)
Measure: Median (95% Confidence Interval); unit: mm
Arm/Group | Benzocaine | Saline Spray
Number analyzed (Participants) | 15 | 15
mm | 50.6 [-7.4 to 98.8] | 70.4 [19.8 to 100]
Statistical Analysis 1: Comparison: Benzocaine vs Saline Spray; An a priori sample size calculation determined at least 28 patients were needed to detect a clinically significant 13 mm difference in pain score (α=0.05, power =0.80) with a standard deviation of 12 mm. Intention to treat analysis was performed; Test type: Superiority or Other; p = 0.43, Wilcoxon (Mann-Whitney); Differences in the median change in pain scores were assessed using Wilcoxon rank sum test

2. Secondary Outcome: Patient Satisfaction
Description: The patient's satisfaction will be assessed using a validated satisfaction scale 30 minutes post procedure.
Time Frame: 30 minutes post procedure
Measure: Number; unit: participants
Arm/Group | Benzocaine | Saline Spray
Number analyzed (Participants) | 15 | 15
participants
  Extremely satisfied | 10 | 10
  Very satisfied | 2 | 4
  Satisfied | 2 | 0
Statistical Analysis 1: Comparison: Benzocaine vs Saline Spray; Fisher exact test was used to assess differences in satisfaction scores by treatment group. Correlation between pain and satisfaction scores was assessed by Spearman's correlation coefficient; Test type: Superiority or Other; p = 0.4, Fisher Exact

3. Secondary Outcome: Change in Pain Score From Pre-procedure to 5 Minutes Post Procedure.
Description: The patients pain scores will also be assessed at 5 minutes post procedure and the change in pain scores from baseline to this time points will be analyzed. The pain scores will be subtracted to obtain the change in pain score
Time Frame: 5 minutes
Measure: Median (95% Confidence Interval); unit: mm
Arm/Group | Benzocaine | Saline Spray
Number analyzed (Participants) | 15 | 15
mm | -11.1 [-90.1 to 18.5] | -37 [-100 to 1.2]
Statistical Analysis 1: Comparison: Benzocaine vs Saline Spray; Test type: Superiority or Other; p = 0.33, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Benzocaine | Saline Spray
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
Standard deviations were wider than anticipated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No